CLINICAL TRIAL: NCT05019937
Title: A Randomized Controlled Trial in Schools Aimed at Testing the Effectiveness of Implementation Strategies, Including Mechanism of Change, on Adherence to the Guideline for the Prevention of Common Mental Disorders at the Workplace.
Brief Title: Exploring Effectiveness and Mechanism of Change of an Implementation Strategy on Guideline Implementation in Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lydia Kwak (Other)
Collaborators: Swedish Council for Working Life and Social Research (Other)
Responsible Party: Sponsor-Investigator, Lydia Kwak, Associate professor, lecturer, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-01214; 2020-01214 (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2021-08-09; First posted 2021-08-25 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Mental Disorder; Stress
Keywords: Guideline; Implementation; Implementation strategies; Mechanism of change; Workplaces; Organisational and social work environment; Schools
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Two-armed cluster-randomized controlled trail
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multifaceted implementation strategy (Experimental): Schools randomized to this arm will be exposed to a multifaceted implementation strategy, which contains five implementation components
  Interventions: Behavioral: Educational meeting; Behavioral: Implementation team; Behavioral: Workshops; Behavioral: Plan-Do-Study-Act improvement cycles; Behavioral: Internal facilitator
- Single implementation strategy (Active Comparator): Schools randomized to this arm will be exposed to a single implementation strategy, which contains one implementation component
  Interventions: Behavioral: Educational meeting

INTERVENTIONS:
Behavioral: Educational meeting — The investigators will hold a full-day educational meeting. The meeting will include educating 4-5 representatives of each school, and school-district representatives about the guideline and the advantages of adhering to the guideline.
  Other Names: Conduct an educational meeting (15) - ERIC cluster Train and educate stakeholders
Behavioral: Implementation team — The school-principal forms an implementation team that is responsible for implementing the guideline within their school. The team members (n=4-5) reflect on the implementation progress, make, and refine plans according to Plan-Do-Study-Act, share lessons learned and support each other.
  Other Names: Organize implementation teams (48) - ERIC cluster Develop stakeholder inter-relationships
  Arms: Multifaceted implementation strategy
Behavioral: Workshops — The investigators will hold 5 workshops. Workshops will include providing in-depth knowledge and skills on the guideline recommendations. During each workshop one of the guideline recommendations will be presented and discussed.
  Moreover, the concept of Plan-Do-Study-Act will be introduced and how it can be used to implement the guideline recommendation(s). During each workshop, the implementation team will share with the group their developed PLAN and barriers and facilitators that have influenced the execution of the PLAN.
  Other Names: Conduct ongoing training (19) - ERIC cluster Train and educate stakeholders
  Arms: Multifaceted implementation strategy
Behavioral: Plan-Do-Study-Act improvement cycles — The implementation team will implement the guideline in a cyclical manner by using Plan-Do-Study-Act. First a Plan is specified during the workshop by using SMART-goals, next the change is carried out between workshops (Do), the implementation team analyses whether it went well and what needs to be improved (Study), changes are made (Act) and finally the next cycle is planned.
  Other Names: Conduct cyclical small tests of change (14) - ERIC cluster Use evaluative and iterative strategies
  Arms: Multifaceted implementation strategy
Behavioral: Internal facilitator — Each municipality assigns one or more internal facilitators, for example HR-strategist. The internal facilitator will meet their local implementation teams during the educational meeting and workshops. Further meeting can be scheduled based on the needs of each implementation team. The internal facilitator will create a supportive environment within which knowledge is exchanged, barriers to implementation identified, and processes or solutions to overcome those barriers developed, applied, and refined. Moreover, the internal facilitator will establish ongoing audit and feedback processes.
  Other Names: Implementation facilitation (10) - ERIC cluster Provide interactive assistance
  Arms: Multifaceted implementation strategy

SUMMARY:
This project is a two-armed randomized-controlled trial exploring the effectiveness and mechanisms of change of two different implementation strategies for implementing the Guideline for the prevention of mental ill-health at the workplace. The project will be conducted among public primary and secondary schools belonging to four municipalities in Sweden. Data will be collected with mixed-methods at baseline and different time-points of follow-up.

DETAILED DESCRIPTION:
There is an urgent need for more knowledge on effective implementation strategies, as two-thirds of implementation efforts fail to achieve the intended change, and half have no effect on outcomes of interest. These implementation failures are partly due to the limited understanding of how implementation strategies work-the mechanisms of change through which implementation strategies affect implementation. This project will fill this research-gap by exploring mechanism of change during a cluster randomized controlled trial that compares the effectiveness of two implementation strategies for implementing the Guideline for the prevention of mental ill-health at the workplace in schools. Schools are chosen as the setting for implementation given the high prevalence of mental ill-health among teachers. Moreover, schools lack a structured approach to the prevention of mental ill-health. The aim of the project is to investigate how implementation strategies affect the defined mechanisms and guideline implementation. Mechanisms that will be tested include hypothesized mediators originating from the individual behavior change theory COM-B. The project will be conducted in public primary and secondary schools in four municipalities in Sweden. Data will be collected with mixed-methods from school-management and personnel at baseline, and different time-points during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* All personnel employed by the school

Exclusion Criteria:

* Personnel not employed by the school (e.g. cleaning- and canteen-personnel)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2276 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Guideline adherence | At baseline, 12- and 24 months follow-up
  Change from baseline in adherence to the recommendations of the guideline during 12-, and 24-months follow-up. Guideline adherence will be assessed with a checklist and questionnaire developed for the purpose of the project.

SECONDARY OUTCOMES:
Self-perceived health | At baseline, 12- and 24-months follow-up
  Change from baseline in self-perceived health during 12-, and 24-months follow-up. Self-perceived health is assessed with a single question from the SF-12 Health Survey (Ware JE, Kosinski MA, & DM, 2002)
Self-reported stress | At baseline, 12- and 24-months follow-up
  Change from baseline in self-reported stress during 12-, and 24-months follow-up. Self-reported stress is assessed with a single item (Arapovic-Johansson, Wahlin, Kwak, Bjorklund, & Jensen, 2017; Elo, Leppanen, & Jahkola, 2003).
Psychosocial safety climate | At baseline, 12- and 24-months follow-up
  Change from baseline in psychosocial safety climate during 12-, and 24-months follow-up. Psychosocial safety climate is assessed with PSC-4, which is a short questionnaire with 4 items measuring the Psychosocial Safety Climate at work (Berthelsen & Muhonen, 2017)
Organisational readiness to implement | At baseline, 12- and 24-months follow-up
  Change from baseline in organisational readiness to implement the guideline during 12-, and 24-months follow-up. Organisational readiness to implement will be assessed with the Leader Readiness to Implement Tool (LRIT) developed and validated by Cook et al. manuscript submitted. With the tool a total readiness index will be calculated, but also a change efficacy score and a change commitment score indicating the confidence and commitment to implement the guideline within the organisation (school).
Implementation leadership | At baseline, 12- and 24-months follow-up
  Change from baseline in implementation leadership during 12- and 24-months follow-up. Implementation leadership will be assessed with items from the S-ILS (Aarons, Ehrhart, & Farahnak, 2014; Lyon et al., 2018). The S-ILS assesses the degree to which a leader is Proactive, Knowledgeable, Supportive, and Perseverant in implementing evidence-based practice (the guideline). Scores for the subscales will be calculated and a total score for the S-ILS is calculated by taking a mean of the scale scores.

OTHER OUTCOMES:
Knowledge | 12-months
  Change in knowledge during 12-months. Knowledge is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for knowledge.
Skills | 12-months
  Change in skills during 12-months. Skills is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for skills.
Social/professional role and identity | 12-months
  Change in social/professional role and identity during 12-months. Social/professional role and identity is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for social/professional role and identity.
Beliefs about capabilities | 12-months
  Change in beliefs about capabilities during 12-months. Beliefs about capabilities is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for beliefs about capabilities.
Beliefs about consequences | 12-months
  Change in beliefs about consequences during 12-months. Beliefs about consequences is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for beliefs about consequences.
Reinforcement | 12-months
  Change in reinforcement during 12-months. Reinforcement is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for reinforcement.
Intentions | 12-months
  Change in intention during 12-months. Intention is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for intention.
Goals | 12-months
  Change in goals during 12-months. Goals is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for goals.
Environmental context and resources | 12-months
  Change in environmental context and resources during 12-months. Environmental context and resources is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for environmental context and resources.
Social influences | 12-months
  Change in social influences during 12-months. Social influences is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for social influences.
Behavioral regulation | 12-months
  Change in behavioral regulation during 12-months. Behavioural regulation is assessed with items from the Theoretical Domains Framework (TDF)-questionnaire (Huijg et al., 2014). The TDF-questionnaire assesses factors influencing the implementation of the guideline. In the project the questionnaire will be used to asses potential mediators that influence guideline implementation. A sum-score will be calculated for behavioural regulation.

CONTACTS AND LOCATIONS:
Overall Officials: Lydia Kwak, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Unit for Intervention and Implementation Research for Worker Health, Institute for Environmental Medicine, Karolinska Institute, Stockholm, Sweden

REFERENCES:
- [Derived] Rodlund A, Toropova A, Lengnick-Hall R, Powell BJ, Schafer Elinder L, Bjorklund C, Kwak L. A cluster-randomized controlled trial assessing the effectiveness of a multifaceted versus a discrete implementation strategy on fidelity to an occupational guideline for the prevention of mental health problems at the workplace: a dual perspective from Swedish schools. Implement Sci Commun. 2025 Nov 21;6(1):127. doi: 10.1186/s43058-025-00821-x. PMID 41272910